CLINICAL TRIAL: NCT01022580
Title: Trial of Late Surfactant for Prevention of Bronchopulmonary Dysplasia: A Study in Ventilated Preterm Infants Receiving Inhaled Nitric Oxide
Brief Title: Trial of Late Surfactant for Prevention of Bronchopulmonary Dysplasia
Acronym: TOLSURF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Roberta Ballard (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Roberta Ballard, Professor of Pediatrics, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H10842-33541-01A; U01HL094338 (NIH)
Record Dates: First submitted 2009-11-19; First posted 2009-12-01 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: nitric oxide; surfactant; BPD; prematurity; neonates; iNO; pulmonary outcome; neurodevelopmental outcome; Infasurf; lung function; Surfactant Dysfunction; Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth; Surfactant Dysfunction | interventions — Therapeutics; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infasurf surfactant (ONY, Inc.) (Active Comparator): Infants already receiving inhaled nitric oxide will receive scheduled doses of late surfactant (Infasurf) on study days 0, 2, 4, 6 and 8.
  Interventions: Drug: Infasurf surfactant (ONY, Inc.)
- Sham (No Treatment) (Sham Comparator): Infants already receiving inhaled nitric oxide will receive "Sham (no treatment)" doses on study days 0,2,4,6, and 8.
  Interventions: Drug: Sham (No Treatment)

INTERVENTIONS:
Drug: Infasurf surfactant (ONY, Inc.) — Late doses of Infasurf 3ml/kg will be given to infants on study days 0, 2, 4, 6 and 8 as long as infant remains intubated.
  Other Names: Treatment
  Arms: Infasurf surfactant (ONY, Inc.)
Drug: Sham (No Treatment) — Late doses of Sham (No treatment) will be given to infants on study days 0, 2, 4, 6 and 8 as long as infant remains intubated.
  Other Names: Control
  Arms: Sham (No Treatment)

SUMMARY:
The purpose of this study is to determine if late doses of Infasurf surfactant given when patients are receiving inhaled nitric oxide will interact to improve surfactant function and increase survival without BPD in treated infants.

DETAILED DESCRIPTION:
This is a multi-center, blinded, randomized controlled clinical trial to evaluate the effects of booster doses of exogenous surfactant (Infasurf®, calfactant) in addition to inhaled nitric oxide (iNO) on the outcome of survival without bronchopulmonary dysplasia (BPD, or chronic lung disease of prematurity, characterized by chronic lung dysfunction) at 36 weeks' post-menstrual age (PMA) in extremely low gestational age (ELGAN) infants that are at high risk of the development of BPD. This multi-center trial, with a planned enrollment of 524 infants, will also enable us to evaluate for any adverse effects of late surfactant treatment on short- and long-term outcomes, as we will be collecting data on effects of dosing of late surfactant, co-morbidities of prematurity and neurodevelopmental and pulmonary outcome at 1 year and 24 months corrected age. In addition, we will collect biological specimens for evaluation of the effects of late surfactant replacement therapy (administered as described in this trial) on surfactant function and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* <=28 0/7 weeks gestational age
* Day of life 7-14
* Intubated and mechanically ventilated
* Plan to treat with inhaled nitric oxide

Exclusion Criteria:

* Serious congenital malformations or chromosomal abnormalities
* Life expectancy <7 days from enrollment
* Clinically unstable
* Less tha 48 hours since last dose surfactant
* Ability to obtain 36 week primary outcome information is unlikely

Ages: 7 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 511 (Actual)
Dates: Start 2010-01; Primary Completion 2013-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberta A Ballard, MD, Principal Investigator — University of California, San Francisco
Locations (21):
- United States (21):
  - University of Arkansas - Arkansas Childrens Hospital, Little Rock, Arkansas
  - Alta Bates Medical Center, Berkeley, California
  - Oakland Children's Hospital, Oakland, California
  - University of California, San Francisco, San Francisco, California
  - Wolfson Children's Hospital and Shands HospitaL, Jacksonville, Florida
  - Florida Hospital for Children, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - Childrens Hospital and Clinics of Minnesota- Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Children's Hospital and Clinics of Minnesota - St Paul, Saint Paul, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Women's and Children's Hospital of Buffalo, Buffalo, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Wake Forest University- Forsyth Hospital and Brenner Hospital, Winston-Salem, North Carolina
  - Medical University of South Carolina(MUSC), Charleston, South Carolina
  - UT Memphis- Memphis Medical Center, Memphis, Tennessee
  - UT Houston Health Science Center, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Washington, Seattle, Seattle, Washington

REFERENCES:
- [Background] Ballard RA, Truog WE, Cnaan A, Martin RJ, Ballard PL, Merrill JD, Walsh MC, Durand DJ, Mayock DE, Eichenwald EC, Null DR, Hudak ML, Puri AR, Golombek SG, Courtney SE, Stewart DL, Welty SE, Phibbs RH, Hibbs AM, Luan X, Wadlinger SR, Asselin JM, Coburn CE; NO CLD Study Group. Inhaled nitric oxide in preterm infants undergoing mechanical ventilation. N Engl J Med. 2006 Jul 27;355(4):343-53. doi: 10.1056/NEJMoa061088. PMID 16870913
- [Background] Ballard PL, Merrill JD, Truog WE, Godinez RI, Godinez MH, McDevitt TM, Ning Y, Golombek SG, Parton LA, Luan X, Cnaan A, Ballard RA. Surfactant function and composition in premature infants treated with inhaled nitric oxide. Pediatrics. 2007 Aug;120(2):346-53. doi: 10.1542/peds.2007-0095. PMID 17671061
- [Background] Truog WE, Ballard PL, Norberg M, Golombek S, Savani RC, Merrill JD, Parton LA, Cnaan A, Luan X, Ballard RA; Nitric Oxide (to Prevent) Chronic Lung Disease Study Investigators. Inflammatory markers and mediators in tracheal fluid of premature infants treated with inhaled nitric oxide. Pediatrics. 2007 Apr;119(4):670-8. doi: 10.1542/peds.2006-2683. PMID 17403837
- [Result] Ballard RA, Keller RL, Black DM, Ballard PL, Merrill JD, Eichenwald EC, Truog WE, Mammel MC, Steinhorn RH, Rogers EE, Ryan RM, Durand DJ, Asselin JM, Bendel CM, Bendel-Stenzel EM, Courtney SE, Dhanireddy R, Hudak ML, Koch FR, Mayock DE, McKay VJ, O'Shea TM, Porta NF, Wadhawan R, Palermo L; TOLSURF Study Group. Randomized Trial of Late Surfactant Treatment in Ventilated Preterm Infants Receiving Inhaled Nitric Oxide. J Pediatr. 2016 Jan;168:23-29.e4. doi: 10.1016/j.jpeds.2015.09.031. Epub 2015 Oct 21. PMID 26500107
- [Result] Wai KC, Hibbs AM, Steurer MA, Black DM, Asselin JM, Eichenwald EC, Ballard PL, Ballard RA, Keller RL; Trial of Late Surfactant (TOLSURF) Study Group. Maternal Black Race and Persistent Wheezing Illness in Former Extremely Low Gestational Age Newborns: Secondary Analysis of a Randomized Trial. J Pediatr. 2018 Jul;198:201-208.e3. doi: 10.1016/j.jpeds.2018.02.032. Epub 2018 Apr 4. PMID 29627188
- [Result] Keller RL, Eichenwald EC, Hibbs AM, Rogers EE, Wai KC, Black DM, Ballard PL, Asselin JM, Truog WE, Merrill JD, Mammel MC, Steinhorn RH, Ryan RM, Durand DJ, Bendel CM, Bendel-Stenzel EM, Courtney SE, Dhanireddy R, Hudak ML, Koch FR, Mayock DE, McKay VJ, Helderman J, Porta NF, Wadhawan R, Palermo L, Ballard RA; TOLSURF Study Group. The Randomized, Controlled Trial of Late Surfactant: Effects on Respiratory Outcomes at 1-Year Corrected Age. J Pediatr. 2017 Apr;183:19-25.e2. doi: 10.1016/j.jpeds.2016.12.059. Epub 2017 Jan 16. PMID 28100402
- [Derived] Wai KC, Keller RL, Lusk LA, Ballard RA, Chan DK; Trial of Late Surfactant (TOLSURF) Study Group. Characteristics of Extremely Low Gestational Age Newborns Undergoing Tracheotomy: A Secondary Analysis of the Trial of Late Surfactant Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2017 Jan 1;143(1):13-19. doi: 10.1001/jamaoto.2016.2428. PMID 27583380

RESULTS

PARTICIPANT FLOW:
Groups:
- Infasurf Surfactant (ONY, Inc.): Infants already receiving inhaled nitric oxide will receive scheduled doses of late surfactant (Infasurf) on study days 0, 2, 4, 6 and 8.
  Infasurf surfactant (ONY, Inc.): Late doses of Infasurf 3ml/kg will be given to infants on study days 0, 2, 4, 6 and 8.
- Sham: Infants already receiving inhaled nitric oxide will not receive additional doses of late surfactant (Infasurf).
Period: Overall Study
Arm/Group | Infasurf Surfactant (ONY, Inc.) | Sham
Started | 252 | 259
Completed | 234 (Survived to discharge) | 237 (Survived to discharge.)
Not Completed | 18 | 22
Not completed — Death | 18 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infasurf Surfactant (ONY, Inc.) | Sham | Total
Number analyzed (Participants) | 252 | 259 | 511
Age, Continuous [Mean (Standard Deviation); unit: weeks]
  Gestational Age Weeks | 25.2 (1.2) | 25.2 (1.2) | 25.2 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 121 | 230
  Male | 143 | 138 | 281
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 33 | 56
  Not Hispanic or Latino | 227 | 225 | 452
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 9 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 99 | 91 | 190
  White | 134 | 157 | 291
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 4 | 2 | 6
Respiratory Severity Score (RSS) - MAP x FiO2 [Mean (Standard Deviation); unit: score on a scale] — Respiratory Severity Score (RSS) equals the mean airway pressure (on ventilator or Nasal CPAP) X fraction of inspired oxygen (FiO2). Range can be 0 - 16, higher scores indicating greater disease severity.
  score on a scale | 3.7 (2.3) | 3.8 (2.2) | 3.75 (3.25)
Birthweight [Mean (Standard Deviation); unit: grams] | 700.1 (173.2) | 702.3 (156.0) | 701 (160)

OUTCOME MEASURES:

1. Primary Outcome: Survival Without BPD at 36 Weeks Post Menstrual Age.
Description: BPD was diagnosed as need for respiratory support with either positive pressure and/or oxygen as evaluated by physiological oxygen/flow reduction.
Time Frame: 36 weeks post menstrual age +/- 1 week
Measure: Count of Participants; unit: Participants
Groups:
- Infasurf Surfactant (ONY, Inc.): Infants already receiving inhaled nitric oxide will receive scheduled doses of late surfactant (Infasurf) on study days 0, and repeated Q24-72 hours as long as infant remains ventilated.
  Infasurf surfactant (ONY, Inc.): Late doses of Infasurf 3ml/kg will be given to infants on study days 0, and repeated Q24-72 hours as long as infant remains ventilated.
- Sham: Infants already receiving inhaled nitric oxide will receive scheduled sham (nothing done) doses of late surfactant (nothing done).
  Sham (nothing done) doses will be given to infants on study days 0,and repeated Q24-72 hours as long as infant remains ventilated.
Arm/Group | Infasurf Surfactant (ONY, Inc.) | Sham
Number analyzed (Participants) | 252 | 259
Participants | 79 | 82
Statistical Analysis 1: Comparison: Infasurf Surfactant (ONY, Inc.) vs Sham; Test type: Superiority or Other; p = 0.89, unadj GEE

2. Secondary Outcome: Survival Without BPD at 40 Weeks
Description: as for outcome 1
Time Frame: 40 weeks PMA +/- 1 week
Population: Infants who were No BPD at 36 wk were imputed to be No BPD at 40 wk. Infants discharged on oxygen without a challenge test were assigned Yes BPD.
Measure: Count of Participants; unit: Participants
Groups:
- Infasurf Surfactant (ONY, Inc.): Infants already receiving inhaled nitric oxide will receive scheduled doses of late surfactant (Infasurf) upon entry into study.
  Repeat Infasurf surfactant (ONY, Inc.) doses will be given to infants still ventilated on study days (+/- 24 hours): 2, 4, 6 and 8.
- Sham: Infants already receiving inhaled nitric oxide will receive Sham (no treatment) upon entry into study.
  Repeat Sham doses will be given to infants still ventilated on study days (+/- 24 hours): 2, 4, 6 and 8.
Arm/Group | Infasurf Surfactant (ONY, Inc.) | Sham
Number analyzed (Participants) | 252 | 259
Participants | 148 | 140
Statistical Analysis 1: Comparison: Infasurf Surfactant (ONY, Inc.) vs Sham; Test type: Superiority or Other; p = 0.33, unadj GEE

3. Secondary Outcome: Respiratory Outcomes of TOLSURF Infants at 1 Year Corrected Age
Description: Evaluation of respiratory outcome through the first 12 months after birth. questionnaires were administered by phone at 3,6,9 and 12 months to determine respiratory resource use (medications, home support, and hospitalization) No Pulmonary Morbidity (NoPM) was reported for infants who had no resource use in any quarter and Persistent PM was reported for infants having resource use in 3 or 4 quarters.
Time Frame: 1 year
Population: Infants who survived to discharge and had data from questionaires available
Measure: Count of Participants; unit: Participants
Groups:
- Infasurf Surfactant (ONY, Inc.): Infants who received inhaled nitric oxide and late doses of surfactant will have respiratory questionaires administered by phone at 3,6,9 and 12 months.
- Sham: Infants who received only inhaled nitric oxide will have respiratory questionaires administered by phone at 3,6,9 and 12 months
Arm/Group | Infasurf Surfactant (ONY, Inc.) | Sham
Number analyzed (Participants) | 208 | 240
Participants
  Home respiratory support | 80 | 118
  No PM | 54 | 47
  Persistent PM | 74 | 75

4. Secondary Outcome: Pulmonary Outcomes Through 2 Years of Age
Description: Evaluation of pulmonary outcome at 24 months of age. Evaluation of persistent wheezing based on reported wheezing during both first and second year of life.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Infasurf Surfactant (ONY, Inc.) | Sham
Number analyzed (Participants) | 203 | 217
Participants | 91 | 98

5. Secondary Outcome: Percentage of Participants With Neurodevelopmental Impairment (NDI) at 2 Years.
Description: At 24 months corrected age, children underwent neuropsychological testing with the Bayley Scales of Infant Development-Third Edition (Bayley-3), and composite cognitive, language, and motor scores were collected as well as subscale scores in receptive and expressive speech and fine and gross motor. Infants with greater than one impairment as identified by testing were classified as having neurodevelopmental impairment.
Time Frame: 2 years
Population: Neurodevelopmental testing occurred with only 322 participants.
Measure: Number; unit: percentage of participants
Arm/Group | Infasurf Surfactant (ONY, Inc.) | Sham
Number analyzed (Participants) | 154 | 168
percentage of participants | 28 | 32

ADVERSE EVENTS:
Arm/Group | Infasurf Surfactant (ONY, Inc.) | Sham (No Treatment)
All-Cause Mortality (participants affected / at risk) | 29/252 | 24/259
Serious Adverse Events (participants affected / at risk) | 29/252 | 24/259
Other Adverse Events (participants affected / at risk) | 141/252 | 153/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infasurf Surfactant (ONY, Inc.) (N=252) | Sham (No Treatment) (N=259)
Death (Investigations) | 29 (29) | 24 (24)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infasurf Surfactant (ONY, Inc.) (N=252) | Sham (No Treatment) (N=259)
IVH New or Worsened (General disorders) | 33 (33) | 35 (35) — Evaluation of new or worsened IVH after enrollment.
PDA Requiring Treatment (Cardiac disorders) | 89 (89) | 95 (95) — Incidence of infants who's PDA worsened to the point of needing treatment.
NEC (Gastrointestinal disorders) | 27 (27) | 24 (24) — Incidence of new or worsened NEC after enrollment.
Sepsis (Infections and infestations) | 141 (141) | 153 (153) — Incidence new episodes of culture proven sepsis after enrollment.
ROP Class 4-5 or surgery (Eye disorders) | 34 (34) | 29 (29)

LIMITATIONS AND CAVEATS:
Possible limitations of the trial: Infants 1) may not have had enough surfactant dysfunction to benefit from replacement; or 2) had irreversible lung damage prior to enrollment; or 3) The dose/frequency of replacement surfactant was inadequate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No